CLINICAL TRIAL: NCT05681637
Title: SpO2 Difference Between Fingers of the Hand During Sequential Desaturation and Step Resaturation
Acronym: StatDynSpO2
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Czech Technical University in Prague (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: NVT01/2022
Record Dates: First submitted 2022-12-10; First posted 2023-01-12 (Actual); Last update posted 2023-03-17 (Actual); Status verified 2023-03

CONDITIONS: Hypoxia; Pulse Oximetry; SpO2
MeSH Terms: conditions — Hypoxia

STUDY DESIGN:
Intervention Model Description: Interventional prospective study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Hypoxia (Experimental): Volunteers sequentially inhale three hypoxic gas mixtures each for 2.5 minute. Every measurement will begin with a two-minute stabilization phase, during which the physiological values of the volunteer will be checked. During the experiment, non-invasive SpO2 measurements will be performed continuously on the individual fingers of volunteer hands throughout the experiment.
  Interventions: Other: Breathing mixtures of O2 and N2 and monitoring SpO2 on each finger

INTERVENTIONS:
Other: Breathing mixtures of O2 and N2 and monitoring SpO2 on each finger — Volunteers sequentially inhale three hypoxic gas mixtures each for 2.5 minute. Every measurement will begin with a two-minute stabilization phase, during which the physiological values of the volunteer will be checked. During the experiment, non-invasive SpO2 measurements will be performed continuously on the individual fingers of volunteer hands throughout the experiment.

SUMMARY:
The aim of the project is to experimentally compare the fingers of the hand in terms of measured concentrations of peripheral blood oxygen saturation (SpO2) in healthy humans during gradual desaturation in the range of 60-100% SpO2 and simultaneously during a step change from the hypoxic phase to the recovery phase (return to physiological values).

DETAILED DESCRIPTION:
The finger sensors of pulse oximeters are most often placed on the middle two fingers of the hand. Although there have been many studies looking at the accuracy of different pulse oximeters or comparing fingers in terms of SpO2. There is no study comparing fingers in terms of SpO2 under hypoxic condition with simultaneous randomization of finger probe placement. At the same time, there is no study that compares SpO2 changes between fingers during a step change in blood oxygen saturation. The data obtained could help to improve the reliability of monitoring physiological parameters with pulse oximeters.

ELIGIBILITY:
Inclusion Criteria:

* Passing the initial examination, which will determine the following data: finger circumference, heart rate, blood pressure and blood oxygen saturation

Exclusion Criteria:

* post-traumatic conditions of the upper limbs affecting the perfusion of the fingers or injuries or skin diseases on the fingers.
* pneumothorax or a condition after cardiovascular surgery.
* anemia, bradycardia, hemoglobinopathy or other diseases of the cardiovascular system, pregnancy, diabetes, hypotension or hypertension.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Estimated)
Dates: Start 2023-01-31 (Actual); Primary Completion 2023-05-20 (Estimated); Study Completion 2023-12-20 (Estimated)

PRIMARY OUTCOMES:
Non-invasive SpO2 measurements will be performed continuously on all individual fingers of left hand of volunteers and then the measured values will be compared between each other. | 1 hour
  The experiment can help determine if it depends on which finger the finger sensor will be placed to measure SpO2. Appropriate finger selection for SpO2 measurements could help to better interpret the measured values and possibly increase the success in diagnosing health events.

SECONDARY OUTCOMES:
Non-invasive Perfusion Index measurements will be performed continuously on all individual fingers of left hand of volunteers and then the measured values will be compared between each other. | 1 hour
  The experiment can help determine if it depends on which finger the finger sensor will be placed to measure perfusion index. Measurement of PI is evaluated during for example surgeries.

CONTACTS AND LOCATIONS:
Overall Officials: Karel Roubik, Professor, Study Director — Czech Technical University
Locations (1):
- Czech Technical University in Prague, Kladno, Czechia

REFERENCES:
- [Background] Rafl J, Kulhanek F, Kudrna P, Ort V, Roubik K. Response time of indirectly accessed gas exchange depends on measurement method. Biomed Tech (Berl). 2018 Nov 27;63(6):647-655. doi: 10.1515/bmt-2017-0070. PMID 28802098